CLINICAL TRIAL: NCT00619320
Title: Reducing HIV: Safer Sex Skill Building in Pregnant Drug Abusing Women
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P60MD002256 (Project 2 15378); P60MD002256 (NIH)
Record Dates: First submitted 2008-02-06; First posted 2008-02-20 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: HIV Infections; Substance Use
Keywords: HIV primary prevention; Health promotion; Health behavior; Risk reduction behavior; Sexual behavior; Safe sex; Women's health; Minority health; Pregnant Women; HIV seronegativity
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders; Health Behavior; Risk Reduction Behavior; Sexual Behavior; Safe Sex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Safer Sex Skill Building (SSB) (Experimental): Safer Sex Skill Building Intervention (SSB) A five session behavioral intervention focused on HIV/STD prevention and safer sex negotiation skills
  Interventions: Behavioral: Safer Sex Skills Building (SSB)
- 2 (Active Comparator): one group session focused on standard HIV/STD education
  Interventions: Behavioral: Safer Sex Skills Building (SSB)

INTERVENTIONS:
Behavioral: Safer Sex Skills Building (SSB) — Test the effectiveness of an intervention for reducing sexual risk factors for HIV infection in two samples of pregnant drug-using women. The intervention, Safer Sex Skills Building (SSB)(El Bassel and Schilling (1991, 1992)), is a manual-driven, gender-specific group intervention delivered by mental health counselors. To date, its effectiveness has not been examined in pregnant, drug using women. The proposed study will examine the effectiveness of the intervention in both drug treatment (RBHA, N = 200) and prenatal care (PCC, N = 200) settings. Using a randomized clinical trial design, the study will compare the five-session SSB group intervention to a one-session standard group HIV Education session (ED). Study hypotheses: that women in the SSB intervention will have better outcomes (e.g., fewer unprotected penetrative sexual behaviors) than women in the control group (ED).
  Other Names: Experimental - Safer Sex Skill Building (5 sessions); Active Comparator - HIV/STD Education (1 session)

SUMMARY:
This study will examine safer sex skills building (SSB), a targeted behavioral HIV prevention and risk reduction group intervention in two samples of pregnant drug abusing women.

DETAILED DESCRIPTION:
"Safer Sex Skills Building" in Pregnant Women: Dace Svikis, (Psychology, Ob-Gyn, Psychiatry) PI, Diane Langhorst (Social Work) and Nichole Karjane, (OB-Gyn) Co-Investigators). This study will focus on increasing Safer Sex Skills development among pregnant women at high risk for HIV infection. The "Safer Sex Skill Building" (SSB) program developed by El Bassel and Schilling (1991, 1992), has demonstrated efficacy in national studies in reducing sexual risk for HIV and other STD transmission. This manual-driven, gender-specific intervention has proven effective in reducing sexual risk behaviors in both methadone maintenance and outpatient drug-free patients. To date, however, the intervention has not been tested with pregnant drug abusing women who may actually be at increased risk if they stop using condoms or continue drug use during pregnancy. This study will examine SSB, a targeted behavioral HIV prevention and risk reduction intervention in two samples of pregnant drug abusing women. Using a 2x2 design, a randomized clinical trial will compare the five-session SSB group intervention to a one-session standard group HIV Education intervention (SE). Study findings will provide benchmark data on the efficacy of SSB for HIV and STD prevention in a diverse sample of pregnant drug abusing women.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older, pregnant
* At prenatal care (PCC) site: screen positive for on T-ACE and TWEAK and/or drug CAGE, report drinking 3 or more drinks on at least one occasion and/or using an illicit drug at least once in the 30 days prior to pregnancy awareness, and report at least one incident of unprotected penetrative (vaginal or anal) intercourse with a male partner within the six months prior to baseline assessment.
* At community treatment (RBHA) site, inclusion criteria are the same except post-partum women (i.e., those who gave birth to a child 2 years of age or less) will also be eligible for study enrollment.

Exclusion Criteria:

Both sites:

* Unable to provide informed consent due to cognitive impairment, psychiatric instability, or language barriers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2008-12; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Number of penetrative unprotected sexual intercourse occasions | baseline, 1 month, 3 months, and 6 months post-randomization follow-up assessment
The proportion of sex episodes involving alcohol or other drugs | baseline, 1 month, 3 months, and 6 months post-randomization follow-up assessment
The proportion of penetrative unprotected sex occasions (of all sex occasions) | baseline, 1 month, 3 months, and 6 months post-randomization follow-up assessment

SECONDARY OUTCOMES:
Perceived self-efficacy to carry out safer sex and the carrying of condoms | baseline, 1 month, 3 months, and 6 months post-randomization follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Dace S Svikis, Ph.D., Principal Investigator — Professor, Department of Psychology, Virginia Commonwealth University
Locations (2):
- United States (2):
  - Richmond Behavioral Health Authority (RBHA), Richmond, Virginia
  - Virginia Commonwealth University, Nelson Womens Health (OB) Clinic, Richmond, Virginia